CLINICAL TRIAL: NCT06201078
Title: Phase II Study - Stereotactic Re-irradiation of Local Recurrences of Prostate Cancer After Radiotherapy - PROSTARE (PROstate Cancer STereotActic REirradiation) Trial
Brief Title: Stereotactic Re-irradiation of Local Recurrences of Prostate Cancer After Radiotherapy
Acronym: PROSTARE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Maria Sklodowska-Curie National Research Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: nio-kb/430-72/23
Record Dates: First submitted 2023-12-29; First posted 2024-01-11 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Local Recurrence of Malignant Tumor of Prostate; Radiotherapy
Keywords: local recurrence; prostate; radiotherapy; salvage
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Salvage SBRT for locally recurrent prostate cancer after radiotherapy (Experimental): SBRT: 5 x 6.75 Gy (every other day) to the total dose of 33.75 Gy
  Interventions: Radiation: Stereotactic Body Radiotherapy

INTERVENTIONS:
Radiation: Stereotactic Body Radiotherapy — Salvage SBRT will be performed in three subgroups of patients with local recurrence:
  Group A - after conventionally fractionated/moderately hypofractionated definitive radiotherapy; Group B - after prostatectomy and postoperative radiotherapy; Group C - after ultrahypofractionated definitive SBRT
  Target volumes:
  GTV- tumour visible on MRI and PET-CT; CTV- 1-3 mm margin around GTV PTV- 3 mm around CTV*
  *- in cases in which very high accuracy and reproducibility of SBRT are ensured, and the margin overlaps the rectum and/or bladder, it is possible to reduce the margin from these organs to 1 mm.
  Dose constrains:
  The criteria for limiting the dose in nearby organs are not well-defined for repeated irradiation - the following doses should be aimed:
  * Maximum rectal dose ≤103% of the prescribed dose (optimal ≤100%)
  * Maximum bladder dose ≤105% of the prescribed dose (optimal ≤103%)
  Dose-volume constrains:
  Rectum:
  • D30% <15Gy
  Bladder:
  • D30% < 15 Gy

SUMMARY:
The goal of this clinical study is to evaluate the toxicity and efficacy of re-irradiation using focal stereotactic body radiotherapy (SBRT) in patients with local recurrence of prostate cancer after definitive or post-operative radiotherapy.

The main question is the tolerance of such treatment, concerning the incidence of Grade ≥ 2 and Grade ≥ 3 GU and GI toxicity. Also the efficacy of SBRT will be measured in terms of Biochemical Control with other secondary endpoints which include: Biochemical Response, Biochemical Failure-Free Survival, Metastases-Free Survival, Relapse-Free Survial, Local Control, Overall Survival and patients' reported tolerance measured with Quality of Life questionnaires (QoL C-30 and PR-25).

The evaluation of the tolerance and effectiveness of stereotactic radiotherapy (SBRT) will be performed in 3 subgroups: in patients with local recurrence after conventionally fractionated/moderately hypofractionated definitive radiotherapy (Group A) or ultrahypofractionated definitive SBRT (Group C) or after prostatectomy and post-operative radiotherapy (Group B).

The study group is planned to include 55 patients.

DETAILED DESCRIPTION:
The diagnosis of local recurrence after radiotherapy in patients with prostate cancer is a serious clinical problem. Interventional salvage treatment in the previously irradiated area is difficult with safety issues of special concern. According to the MASTER meta-analysis the effectiveness of various local salvage methods turned out to be comparable in patients with local recurrence after definitive radiotherapy. Stereotactic radiotherapy (SBRT) had the best toxicity profile, so this non-invasive treatment may be a suitable alternative to other methods. A particular problem is local recurrences after post-prostatectomy radiotherapy. The data on SBRT in such setting are even more scarce than in the case of relapses after definitive radiotherapy. Still, they show a low percentage of serious adverse events of grade ≥3 and good treatment tolerance.

Considering the own experience with re-irradiation of patients with prostate cancer, it was decided that re-irradiation should be carried out in the form of focal SBRT. With the objective of enhancing the safety and quality of salvage re-irradiation, and a comprehensive evaluation of the efficacy of this treatment it was determined that it should be implemented as a prospective phase II study- PROSTARE (PROstate cancer STereotActic Reirradiation).

The evaluation of the tolerance and effectiveness of stereotactic radiotherapy (SBRT) will be performed in patients with local recurrence after conventionally fractionated/moderately hypofractionated definitive radiotherapy (Group A), ultrahypofractionated definitive SBRT (Group C), or after prostatectomy and postoperative radiotherapy (Group B).

The study will be conducted as a single-centre study. The evaluation of the safety and effectiveness of such treatment could help develop qualification criteria for repeated irradiation. As a consequence, this should allow for the implementation of this form of treatment into radiotherapy protocols and then, in a controlled and safe way, into clinical practice.

The total sample size will comprise 55 patients. The expected recruitment period is 6 years (10 patients per year).

Requirements for reirradiation with SBRT:

1. Both PET-PSMA and MR of the prostate or prostate bed are required in patients with recurrence after definitive radiotherapy or surgery followed by radiotherapy
2. Fiducial implantation is not routinely required
3. Empty rectum and partially empty/partially filled bladder (improved reproducibility)* during treatment planning and during each fraction of stereotactic radiotherapy
4. Treatment with a linear accelerator is preferred
5. CBCT must be performed before each fraction of SBRT with verification for tumour location (GTV)**
6. Focal radiotherapy, i.e., irradiation of only the visible tumour with an appropriate margin
7. Hormonal treatment is not routinely recommended (according to the ESTRO ACROP consensus) - up to the decision of the attending physician

   * Principles of preparation with laxatives - Bisacodyl is advocated 4-5 hours before SBRT. If the diameter of the rectum on the CT for treatment planning exceeds 4 cm in diameter, the procedure should be repeated after appropriate preparation of the patient.

     * If stereotactic radiotherapy is conducted on the CyberKnife - KV imaging and Tracking verification are required; additionally an assessment of bladder filling in ultrasonography should be performed

ELIGIBILITY:
Inclusion Criteria:

1. Local recurrence of prostate cancer after definitive radiotherapy

   1. biopsy proven or/and
   2. Consistent MRI and PET-PSMA results and PSA growth dynamics
2. Time since primary radiotherapy - at least 2 years
3. Good performance status (ZUBROD 0-1)

   * If the results of the MRI and PET PSMA are inconsistent, and if there is no technical possibility of performing an MRI biopsy, the treatment is acceptable, but repeated imaging (PET or MRI) should be performed to assess the dynamics of the recurrence.

Exclusion Criteria:

1. Polymetastatic dissemination in distant or regional lymph nodes (N1, M1) or oligometastatic dissemination, but not eligible for local forms of metastasis directed therapy (MDT)
2. Tumour volume (GTV) > 14 cc
3. Poor tolerability of primary radiotherapy (≥G3 toxicity) or persistent late toxicity ≥G2 interfering with re-irradiation
4. Severe dysuria before repeated SBRT (e.g., IPSS ≥19)
5. Diseases of the distal part of the rectum or anal canal that may affect SBRT tolerance (e.g., anal fissure)
6. Previous prostate brachytherapy
7. Substantial risk for further urologic interventions (e.g., TURB/TURP)

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2023-07-31 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Tolerance of salvage SBRT | 3 months post-SBRT, 2-years post-SBRT
  Assessment of early and late radiation toxicity: Grade ≥ 3 radiation-induced bladder/urethral (GU) and bowel/rectal (GI) adverse events toxicity or other, according to CTCAE criteria

SECONDARY OUTCOMES:
Tolerance of salvage SBRT | 3 months post-SBRT, every 6 months post SBRT up to 3-years post-SBRT
  Rate of moderate or worse early and late radiation toxicity: Grade ≥ 2 radiation-induced bladder/urethral (GU) and bowel/rectal (GI) adverse events toxicity or other, according to CTCAE criteria
Biochemical Control | 3 months post-SBRT, 6 months post SBRT, every 6 months thereafter up to 5-years post-SBRT
  Biochemical Control will be defined as observations without biochemical recurrence defined as PSA concentration: a. >2 ng/mL above the nadir (according to Phoenix) for groups A and C b. >0.2 ng/ml (according to AUA) for group B
Biochemical Response | 3 months post-SBRT, 6 months post-SBRT, every 6 moths thereafter up to 5-years post-SBRT
  Decrease in PSA level below baseline (pre-SBRT)
Biochemical Failure-Free Survival (BFS) | 3 months post-SBRT, 6 months post SBRT, every 6 months thereafter up to 5-years post-SBRT
  Biochemical Failure Free Survival (BFS) is defined as the time interval between SBRT and biochemical, local, regional failure, distant metastasis or death irrespective of the cause
Metastases-Free Survival | 1-year post SBRT, then annually up to 5-years post-SBRT
  Metastases-Free Survival is the time interval between SBRT and occurrence of distant metastases or death irrespective of the cause
Relapse-Free Survival | 1-year post SBRT, then annually up to 5-years post-SBRT
  Relapse-Free Survival is the time interval between SBRT and occurrence of clinical relapse: local recurrence, regional or distant metastases, start of hormonal therapy, or death irrespective of the cause
Local Control | 1-year post SBRT, then annually up to 5-years post-SBRT
  Local Control is defined as the observations without local failure (within prostate or prostate bed):
  1. in-field
  2. out-field
Overall Surival | 3 months post-SBRT, 6 months post-SBRT, every 6 moths thereafter up to 5-years post-SBRT
  Overall Survival is the time interval between SBRT and patient death irrespective of the cause
Patients' reported Quality of Life | 2-years post SBRT, 3-years post SBRT
  Evaluation of EORTC QLQ-C30 and PR-25 questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Wojciech Majewski, MD, PhD, Principal Investigator — Maria Sklodowska Curie Memorial Research Institute of Oncology
Locations (1):
- Maria Sklodowska Memorial Research Institute of Oncology, Gliwice, Poland

REFERENCES:
- [Background] Valle LF, Lehrer EJ, Markovic D, Elashoff D, Levin-Epstein R, Karnes RJ, Reiter RE, Rettig M, Calais J, Nickols NG, Dess RT, Spratt DE, Steinberg ML, Nguyen PL, Davis BJ, Zaorsky NG, Kishan AU. A Systematic Review and Meta-analysis of Local Salvage Therapies After Radiotherapy for Prostate Cancer (MASTER). Eur Urol. 2021 Sep;80(3):280-292. doi: 10.1016/j.eururo.2020.11.010. Epub 2020 Dec 11. PMID 33309278
- [Background] Miszczyk M, Kraszkiewicz M, Moll M, Kaminiow K, Sobel S, Dolla L, Wojcieszek P, Rajwa P, Yanagisawa T, Nowicka Z, Shariat SF, Goldner G, Miszczyk L, Majewski W. Long-Term Outcomes of Stereotactic Body Radiotherapy (SBRT) for Intraprostatic Relapse after Definitive Radiotherapy for Prostate Cancer: Patterns of Failure and Association between Volume of Irradiation and Late Toxicity. Cancers (Basel). 2023 Feb 13;15(4):1180. doi: 10.3390/cancers15041180. PMID 36831523
- [Background] Jereczek-Fossa BA, Marvaso G, Zaffaroni M, Gugliandolo SG, Zerini D, Corso F, Gandini S, Alongi F, Bossi A, Cornford P, De Bari B, Fonteyne V, Hoskin P, Pieters BR, Tree AC, Arcangeli S, Fuller DB, Franzese C, Hannoun-Levi JM, Janoray G, Kerkmeijer L, Kwok Y, Livi L, Loi M, Miralbell R, Pasquier D, Pinkawa M, Scher N, Scorsetti M, Shelan M, Toledano A, van As N, Vavassori A, Zilli T, Pepa M, Ost P; on the behalf of the European Society for Radiotherapy, Oncology Advisory Committee on Radiation Oncology Practice (ESTRO ACROP). Salvage stereotactic body radiotherapy (SBRT) for intraprostatic relapse after prostate cancer radiotherapy: An ESTRO ACROP Delphi consensus. Cancer Treat Rev. 2021 Jul;98:102206. doi: 10.1016/j.ctrv.2021.102206. Epub 2021 Apr 20. PMID 33965893
- [Background] Archer P, Marvaso G, Detti B, Colombo F, Francolini G, Vandendorpe B, Thananayagam MA, Baty M, De Crevoisier R, Alongi F, Nicosia L, Scher N, Toledano A, Di Muzio N, Fodor A, Zilli T, Franzese C, Scorsetti M, Shelan M, Triggiani L, Aymes E, Le Deley MC, Jereczek-Fossa BA, Pasquier D. Salvage Stereotactic Reirradiation for Local Recurrence in the Prostatic Bed After Prostatectomy: A Retrospective Multicenter Study. Eur Urol Oncol. 2023 Jun;6(3):303-310. doi: 10.1016/j.euo.2023.03.005. Epub 2023 Apr 1. PMID 37012102
- [Background] Schroder C, Tang H, Windisch P, Zwahlen DR, Buchali A, Vu E, Bostel T, Sprave T, Zilli T, Murthy V, Forster R. Stereotactic Radiotherapy after Radical Prostatectomy in Patients with Prostate Cancer in the Adjuvant or Salvage Setting: A Systematic Review. Cancers (Basel). 2022 Jan 29;14(3):696. doi: 10.3390/cancers14030696. PMID 35158961